CLINICAL TRIAL: NCT00173823
Title: Malnutrition and Inflammation in Taiwan: Prospective Outcome Evaluation Method (MIT-POEM) in Dialysis Patients
Brief Title: Malnutrition and Inflammation in Dialysis Patients in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700840
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2006-03-13 (Estimated); Status verified 2005-08

CONDITIONS: Hemodialysis; Hypercholesterolemia; Malnutrition; Inflammation; Kidney Failure, Chronic
MeSH Terms: conditions — Hypercholesterolemia; Malnutrition; Inflammation; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
According to the reports of the United States Renal Data System (USRDS), there is a 25% annual mortality rate with nearly 50% of all reported maintenance hemodialysis (HD) patient deaths attributed to atherosclerosis-related complications. Although traditional risk factors of cardiovascular disease (CVD) are common in end-stage renal disease (ESRD) patients, they alone may be insufficient to account for their high prevalence of CVD. Recent evidence demonstrated high plasma homocysteine levels have been established as a risk factor of chronic inflammation and atherosclerosis in patients with ESRD.

Malnutrition and inflammation was associated with poor quality of life, morbidity and mortality. We, the researchers at National Taiwan University Hospital, hope to establish the best predictive profile of HD patient outcome. Thus, we establish several protocols to complete this work.

ELIGIBILITY:
Inclusion Criteria:

* On HD three times a week for more than 3 months (minimizing the confounding effects of residual renal function)

Exclusion Criteria:

* Malignancy;
* Obvious infections or inflammatory diseases;
* Preexisting haematological disorders; and,
* Clinically significant bleeding, transfusion, hospitalization, surgery, or renal transplantation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500
Dates: Start 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Kang Chiang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital and collegues, Taipei, Taiwan